CLINICAL TRIAL: NCT04665271
Title: Acceptability and Efficacy of Zemedy App Versus Education and Relaxation Training App for IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Bold Health Inc. (Industry)
Responsible Party: Principal Investigator, Melissa Hunt, PhD, Associate Director of Clinical Training, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 844160
Record Dates: First submitted 2020-11-12; First posted 2020-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: cognitive behavioral therapy
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Active control with cross-over at post-treatment and three month follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment - Zemedy App (Experimental): Participants will be given immediate access to the Zemedy app for IBS.
  Interventions: Behavioral: Zemedy App
- Active Control - Education and Relaxation Training App (Active Comparator): Participants will be given access to a education and relaxation training app. After 8 weeks they will then be crossed over to the Zemedy app.
  Interventions: Behavioral: Zemedy App

INTERVENTIONS:
Behavioral: Zemedy App — Digital smart phone app that delivers cognitive-behavioral therapy for IBS

SUMMARY:
The purpose of this research is to assess if a new digital app version of a self-help intervention for Irritable Bowel Syndrome (IBS), is an acceptable and effective treatment for improving the overall quality of life in patients with IBS.

DETAILED DESCRIPTION:
The aim of the current study is to test the acceptability and efficacy of an updated digital app for IBS patients. The design of the study is experimental. There will be two experimental groups, an immediate treatment group and an active control group. Once consented and enrolled, participants will be randomly assigned to either the immediate treatment group or the active control group by the coin toss feature of random.org. Participants in the immediate treatment group will be able to download the app at no cost. Participants in the control group will be given access to an education and relaxation training control app at no cost to them. At 8 weeks after enrollment, all participants in both groups will receive a battery of follow-up questionnaires (the same that they answered directly after consenting in the beginning of the study as baseline measures). Upon receipt of the 8 week questionnaire data, participants in the control group will be given access to the Zemedy app. After having had access to the app for 8 weeks, control participants will be asked to complete another set of questionnaires. All participants will receive 3 month post-treatment follow-up questionnaires. The research method is experimental, cross over (randomized controlled trial) with a control control. Participation in the study will last approximately 4.5 months, depending on the subjects willingness to participate and rate of completion.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of physician diagnosis of IBS.
* At least 18 years of age.

Exclusion Criteria:

* Severe depression or suicidality
* Comorbid GI disorder such as inflammatory bowel disease or celiac disease.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Quality of Life (IBSQoL) | 8 weeks
  IBS specific health related quality of life measure. Scale scores range from 0-100 with higher scores reflecting more impairment (worse outcome)
Gastrointestinal Symptom Rating Scale (GSRS) | 8 weeks
  Gastrointestinal Symptom Rating Scale. Scale scores range from 0-78 with high scores representing worse GI symptoms.

SECONDARY OUTCOMES:
GI-Cognitions Questionnaire (GICog) | 8 weeks
  Scale measures distorted, catastrophic beliefs about the social and occupational implications of having gastrointestinal symptoms. Scale scores range from 0 to 64 with higher scores representing worse outcomes (more distorted, catastrophic beliefs about GI symptoms)
Visceral Sensitivity Index (VSI) | 8 weeks
  Scale measures anxiety about visceral (gut) sensations. Scale scores range from 0 to 75 with higher scores representing more anxiety.
Fear of Food Questionnaire (FFQ) | 8 weeks
  Scale measures fear of food and aversive consequences of eating. Scale scores range from 0-90 with higher scores representing more fear and impairment.
Beck Depression Inventory (BDI) | 8 weeks
  Measures depressive symptoms. Scale scores range from 0 to 63 with higher scores representing more severe depressive symptoms.
Work Productivity and Activity Impairment (WPAI) | 8 weeks
  Measures occupational impairment stemming from a health condition. scores range from 0 to 30 with higher scores representing more impairment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hunt MG, Dalvie A, Ipek S, Wasman B. Acceptability and efficacy of the Zemedy app versus a relaxation training and meditation app for IBS: protocol for a randomised controlled trial. BMJ Open. 2022 Jan 17;12(1):e055014. doi: 10.1136/bmjopen-2021-055014. PMID 35039299

DOCUMENTS (3):
  • Study Protocol (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT04665271/Prot_001.pdf
  • Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT04665271/SAP_002.pdf
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT04665271/ICF_000.pdf